CLINICAL TRIAL: NCT03539393
Title: Fremanezumab (TEV-48125) Compassionate Use Program for Pediatric Patients (6 to 17 Years) With Chronic or Episodic Migraine
Brief Title: Fremanezumab Compassionate Use Program for Pediatric Patients
Status: Available | Type: Expanded Access
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TV48125-CNS-80005; TV48125-MH-80011 (Other: Sponsor)
Record Dates: First submitted 2018-05-15; First posted 2018-05-29 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — fremanezumab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Fremanezumab — For patients who enter this program, the monthly dose of fremanezumab to be administered will be confirmed or adjusted, as appropriate, based on the patient's weight every 3 months.
  Other Names: TEV-48125

SUMMARY:
This is a Compassionate Use Program (CUP) based on a licensed physician's unsolicited request. Specifically, this CUP is for male and female pediatric patients 6 to 17 years with a diagnosis of either episodic or chronic migraine who have successfully completed the Teva sponsored study TV48125-CNS-30084 (SPACE study).

DETAILED DESCRIPTION:
Patients must have successfully completed the clinical trial according to the 30084 protocol, without any major protocol violations or tolerability issues, or who are anticipated to complete this trial within the next 2months, and whose Requesting/Treating Physician is requesting continued supply of the investigational medicinal product (IMP) known as TEV-48125 (fremanezumab) on behalf of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients may enter this CUP after successfully completing TV48125-CNS-30084 and all End of Study procedures
* In the opinion of your physician/investigator are able to continue IMP (fremanezumab) in a safe and compliant way.

Exclusion Criteria:

* Additional criteria may apply, please contact your physician/investigator for more information.

Ages: 6 Years to 17 Years | Sex: All
Age Groups: Child